CLINICAL TRIAL: NCT02982057
Title: A Randomized Trial of the Treatment of Non- Culprit Lesion After STEMI: Bioresorbable Vascular Scaffold Versus Optimal Medical Therapy (NCLstudy)
Brief Title: Non Culprit Lesion Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Non Culprit Lesion Study
Record Dates: First submitted 2016-11-07; First posted 2016-12-05 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bioresorbable vascular scaffold(BVS)+ OMT (Active Comparator): hypothesis: scaffolding a non culprit coronary plaque with BVS could facilitate the stabilization process into the atherosclerotic plaque with modification of plaque morphology.
  Intervention:Device
  Interventions: Device: the ABSORB:bioresorbable vascular scaffold
- OMT (Active Comparator): Comparator with ONLY optimal medical treatment (OMT): the aim of the study is to compare the evolution of non culprit lesions after treatment by BVS versus Optimal Medical Therapy at 2 years follow- up.
  Intervention: medical treatment
  Interventions: Drug: O.M.T

INTERVENTIONS:
Device: the ABSORB:bioresorbable vascular scaffold
  Other Names: to compare to optimal medical treatment
  Arms: Bioresorbable vascular scaffold(BVS)+ OMT
Drug: O.M.T
  Other Names: to compare with device
  Arms: OMT

SUMMARY:
The aim of the present study is to compare the evolution of non culprit lesions after treatment by BVS versus optimal medical therapy at 2-years follow- up

DETAILED DESCRIPTION:
Objectives and hypothesis: scaffolding a non culprit /vulnerable coronary plaque with BVS could facilitate the stabilization process into the atherosclerotic plaque with modifications of plaque morphology, especially the lipid content which is considered as one of the main factor leading to recurrent MACE after an ACS.

The interaction between the polymer Platform and the vessel wall, the effect of the everolimus on neointima growth and cellular response into the media could reduce the inflammatory process into the vulnerable plaque could be different Under OMT and BVS implantation.

ELIGIBILITY:
Inclusion Criteria:

* STEMI and multivessel ASCL
* Successful and uneventful primary PCI
* Non culprit lesion > /= 2.5mm RVD suitable for investigation by FFR
* At least one segment of minimum 10 mm length containing a non culprit lesion

Exclusion Criteria:

* non compliant profile
* patient not able to sign an IC
* cardiogenic shock
* left main disease
* GFR<30ml/min/m2
* previous CABG
* LVEF<35%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
measure size of the vulnerable plaque | 2 years
  the size of the vulnerable plaque measured by angio FU at 2 years with an investigation of the same segment than at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- StLuc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes